CLINICAL TRIAL: NCT06004986
Title: DUPI REDUCE Trial (DUPIlumab Dose REDUCtion in Patients With Controlled Atopic Eczema): a Multicenter, Low-intervention, Non-inferiority Randomized Controlled Trial, Embedded in the TREAT NL Registry
Brief Title: DUPIlumab Dose REDUCtion in Patients With Controlled Atopic Eczema
Acronym: DUPI REDUCE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other); Prothya Biosolutions (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Phyllis I. Spuls, Prof. Dr. P.I. Spuls, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-504171-24-00
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema
Keywords: Dupilumab
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dupilumab 300 mg q2w (Active Comparator): Dupilumab s.c. 300 mg every 2 weeks for 24 weeks.
  Interventions: Drug: Dupilumab
- Dupilumab 300 mg q3w (Experimental): Dupilumab s.c. 300 mg every 3 weeks for 24 weeks.
  Interventions: Drug: Dupilumab
- Dupilumab 300 mg q4w (Experimental): Dupilumab s.c. 300 mg every 4 weeks for 24 weeks.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Administering Dupilumab 300 mg at different dosing intervals.
  Other Names: Dupixent

SUMMARY:
The goal of this randomized controlled trial is to study the (cost)effectiveness of extending the intervals between dupilumab doses in patients with well-controlled atopic eczema, while considering physician- and patient-reported disease severity, quality of life, and dupilumab serum trough levels. Patients will be divided randomly into three groups, receiving dupilumab 300 mg every 2 weeks, every 3 weeks, or every 4 weeks. Researchers will then compare the outcomes among these three groups.

DETAILED DESCRIPTION:
While dupilumab is an effective treatment for atopic eczema, it is expensive and not without the risk of unwanted adverse events. Aiming for the lowest possible dose is important. The currently approved dose is a single loading dose of 600 mg, followed by 300 mg every 2 weeks. However, there is evidence that the intervals between doses could be extended in disease-controlled patients while maintaining the same effectiveness. The objective of this study is to assess the (cost)effectiveness and safety of dupilumab dose reduction in patients with controlled atopic eczema. A multicenter, single-blinded, non-inferiority randomized controlled trial will be performed, that is embedded in the TREatment of ATopic eczema (TREAT) NL registry. Adult patients who are already undergoing dupilumab treatment and meet the Treat-to-Target criteria will be assigned randomly to one of three groups: receiving dupilumab 300 mg every 2 weeks, every 3 weeks, or every 4 weeks. The study will cover a duration of 24 weeks, during which participants will have three hospital visits (at week 0, week 16 and week 24) and one telephone appointment (at week 8). These sessions will involve assessments of both physician and patient-reported disease severity, quality of life and the evaluation of dupilumab serum trough levels. Please refer below for a comprehensive overview of the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an adult,
* Has a diagnosis of AE,
* Receives dupilumab 300 mg q2w for the treatment of AE,
* Has controlled disease according to the Treat-to-Target criteria,
* Agrees to the possibility that the dosage of dupilumab will be lowered,
* Has voluntarily signed and dated an informed consent prior to any study related procedure.

Exclusion Criteria:

* The subjects uses or initiates another systemic immunomodulating therapy for AE or another diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean EASI | 24 weeks
  The mean EASI (Eczema Area and Severity Index). The EASI can range from 0 to 72, where a lower score indicates a better outcome.

SECONDARY OUTCOMES:
EASI | 16 weeks
  The mean EASI (Eczema Area and Severity Index). The EASI can range from 0 to 72, where a lower score indicates a better outcome.
vIGA-AD | 16 and 24 weeks
  The mean Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD). The vIGA-AD can range from 0 to 4, where a lower score indicates a better outcome.
PtGA | 16 and 24 weeks
  The mean patient self-reported Global Assessment of disease severity (PtGA). The PtGA can range from 0 to 4, where a lower score indicates a better outcome.
NRS | 16 and 24 weeks
  The mean Peak Pruritus Numerical Rating Scale (NRS). The NRS can range from 0 to 10, where a lower score indicates a better outcome.
POEM | 16 and 24 weeks
  The mean Patient-Oriented Eczema Measure (POEM). The POEM can range from 0 to 28, where a lower score indicates a better outcome.
DLQI | 16 and 24 weeks
  The mean Dermatology Life Quality Index (DLQI). The DLQI can range from 0 to 30, where a lower score indicates a better outcome.
RECAP | 16 and 24 weeks
  The mean Recap of atopic eczema (RECAP). The RECAP can range from 0 to 28, where a lower score indicates a better outcome.
EQ-5D-5L | 16 and 24 weeks
  The mean EuroQol-5 dimensions-5 level/Youth (EQ-5D-5L): adults and caregivers. The EQ-5D-5L can range from 0 to 1, where a higher score indicates a better outcome.
Adapted iMCQ | 16 and 24 weeks
  Adapted iMTA Medical Consumption Questionnaire
Adapted iPCQ | 16 and 24 weeks
  Adapted iMTA Productivity Cost Questionnaire
Adapted iVICQ | 16 and 24 weeks
  Adapted iMTA Valuation of Informal Care Questionnaire
Dupilumab serum trough levels | 0 and 24 weeks
  Dupilumab serum trough levels of 40 patients (n=20 in both the q3w and q4w arms)
Adverse events | 16 and 24 weeks
  Number of adverse events of special interests (AEoSIs), severe adverse events, serious adverse events and suspected unexpected serious adverse reactions (SUSARs), categorized according to medical dictionary for regulatory activities (MedDRA)

CONTACTS AND LOCATIONS:
Overall Officials: Louise AA Gerbens, MD PhD, Study Chair — Amsterdam University Medical Centers; Phyllis I Spuls, MD PhD, Principal Investigator — Amsterdam University Medical Centers; DirkJan Hijnen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Amsterdam University Medical Centers, Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No